CLINICAL TRIAL: NCT05079815
Title: Evaluating the Arabic Version of Aberdeen Menorrhagia Severity Scale (AMSS) for Prediction of Iron Deficiency/ Iron Deficiency Anemia in Women With the Symptom of Chronic Heavy Menstrual Bleeding (HMB)
Brief Title: Heavy Menstrual Bleeding and Iron Deficiency Anemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebraam Faiez Riad, doctor, Assiut University
Other Study IDs: heavy menstrual bleeding
Record Dates: First submitted 2021-10-03; First posted 2021-10-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CBC and serum ferritin — take blood sample for CBC and serum ferritin

SUMMARY:
In the present study, we test the ability of AMSS as a simple tool to identify women with HMB who have ID/ IDA. We will compare the AMSS score to patients' hemoglobin and serum ferritin in women with self-reported HMB and women with normal menstrual flow.

DETAILED DESCRIPTION:
Anemia remains a critical health burden in low- and middle-income countries (LMICs) and a paradigm shift is needed to effectively reduce the prevalence in women. The reproductive years place women at high risk of anemia in general, and iron deficiency anemia (IDA) in particular, largely because of menstrual and delivery -associated blood loss, as the lost iron is often not adequately replenished from dietary sources. Iron deficiency, even without anemia, has profound adverse effects on multiple cellular and metabolic parameters and frequently manifests with impaired cognitive and physical function. In Africa and Eastern Mediterranean regions, around 39% of non-pregnant women and 40-45% of pregnant women have anemia as estimated by The World Health Organization (WHO). Maternal anemia is a risk factor for preterm labor and both maternal and neonatal morbidity and mortality. Although data is limited, 5-28% of women in LMICs experience abnormal uterine bleeding (AUB) yet the importance of menstrual blood loss as an indicator of and a risk factor for anemia is frequently ignored in anemia control and prevention strategies. The condition is further complicated by the fact that both women and their physicians tend to normalize menstrual symptoms. To enable development of comprehensive interventions to address IDA among women in our locality, it is critical to characterize heavy menstrual bleeding (HMB) and its relationship with IDA among women and determine ways to use these data to direct women at risk for IDA to appropriate healthcare services for evaluation and treatment.

For women with HMB, early diagnosis and treatment of anemia is important to prevent its negative health consequences. However, in low resource settings, laboratory facilities are not always available. In addition, laboratory tests may be expensive limiting their use in such circumstances. For this reason, a cheap, simple to use tool to identify women at high risk of anemia who require further evaluation and treatment is needed.

The Aberdeen Menorrhagia Severity Scale (AMSS) is a multi-dimensional scale. It measures quality of life in women with HMB in addition to menstrual bleeding characteristics. AMSS consists of 13 questions. with a 4-point answer to each question. Maximum score is 47, which is converted to a percentage. The lower the scale is associated with better quality of life. The AMSS has been validated against the SF-36, which is a generic scale for measurement of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age women, above age of 18 years old.

Exclusion Criteria:

* women with amenorrhea, postmenopausal women, current or past (in last 6 months) users of hormonal contraceptives, women who have delivered in the past year, or breast fed in past 6 months are all excluded from the study

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — gynaecological research about heavy menstrual bleeding
Study Population: Details on the research will be explained to potentially eligible women. They will be given patient's information leaflet in Arabic (attached). The research team will emphasize that participation in the study is completely voluntary, and women can withdraw at any time without affecting level of care that is provided for them. Eligible women who accept to participate in the study will sign informed consent. Women will be assured on confidentiality and that data will be coded, with no names/ identifying information, and will be kept on a secure server through RedCap operated by Assiut Faculty of Medicine.3.4. Informed consent.
  Consent will be provided
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluating the Arabic version of Aberdeen Menorrhagia Severity Scale (AMSS) for prediction of iron deficiency/ iron deficiency anemia in women with the symptom of chronic heavy menstrual bleeding (HMB) | baseline
  heavy menstrual bleeding and its relation to iron deficiency /iron deficiency anemia

REFERENCES:
- [Background] Cooke AG, McCavit TL, Buchanan GR, Powers JM. Iron Deficiency Anemia in Adolescents Who Present with Heavy Menstrual Bleeding. J Pediatr Adolesc Gynecol. 2017 Apr;30(2):247-250. doi: 10.1016/j.jpag.2016.10.010. Epub 2016 Oct 24. PMID 27789349
- [Background] Peuranpaa P, Heliovaara-Peippo S, Fraser I, Paavonen J, Hurskainen R. Effects of anemia and iron deficiency on quality of life in women with heavy menstrual bleeding. Acta Obstet Gynecol Scand. 2014 Jul;93(7):654-60. doi: 10.1111/aogs.12394. Epub 2014 Jun 9. PMID 24912842